CLINICAL TRIAL: NCT04606082
Title: Intra Uterine Injection of Human Chorionic Gonadotropin Versus Granulocyte Colony Stimulating Factor at Ovum Pick up Day Significantly Increase Implantation Rate and Pregnancy Rate in Intra Cytoplasmic Sperm Injection
Brief Title: Human Chorionic Gonadotropin Versus Granulocyte Colony Stimulating Factor in Increasing Pregnancy Rate in ICSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Elsayed Eldesouky, Assistant professor of obstetrics and gynecology faculty of medicine Alazhar university Cairo, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gyne_415
Record Dates: First submitted 2020-10-23; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Fertility Disorders
MeSH Terms: interventions — Filgrastim; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Granulocyte Colony Stimulated Factor was intrauterine injected once at ovum pick up day
  Interventions: Drug: Granulocyte Colony Stimulated Factor
- Group 2 (Active Comparator): 500 IU Human Chorionic Gonadotropins was injected intrauterine once at ovum pick up day
  Interventions: Drug: Human Chorionic Gonadotropins

INTERVENTIONS:
Drug: Granulocyte Colony Stimulated Factor — GCSF was intrauterine injected once at ovum pick up day
  Other Names: GCSF, Neupogen, Granix and Zarxio
  Arms: Group 1
Drug: Human Chorionic Gonadotropins — 500 IU of HCG was injected intrauterine once at ovum pick up day
  Other Names: HCG, Novarel, and Pregnyl
  Arms: Group 2

SUMMARY:
Intrauterine Granulocyte colony stimulating factor (GCSF) was compared with intrauterine Human Chorionic Gonadotropin (HCG) in increasing clinical pregnancy rate as a primary outcome and ultrasound imaging of gestational sac as a secondary outcome.

DETAILED DESCRIPTION:
Two hundred females with history of recurrent implantation failure and undergoing Intracytoplasmic Sprem injection (ICSI) were randomized into two groups; the first group (100 patients) received intrauterine Granulocyte colony stimulating factor (GCSF) and the second group (100) received intrauterine Human Chorionic Gonadotropin (HCG) at ovum pick up day. The clinical pregnancy rate was evaluated as a primary outcome after 14 days and ultrasound imaging of gestational sac was evaluated as a secondary outcome after 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Females suffering from recurrent implantation failure and undergoing ICSI

Exclusion Criteria:

* presence of comorbidity as diabetes, hypertension, heart diseases, or endocrine disorders

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-30 (Estimated); Primary Completion 2021-01-10 (Estimated); Study Completion 2021-01-10 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | after 14 days from positive pregnancy test
  Clinical pregnancy was evaluated by high HCG levels

SECONDARY OUTCOMES:
Gestational sac imaging | 6 weeks of pregnancy
  ultrasound imaging of Gestational sac after 6 weeks of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Elsayed Eldesouky, Principal Investigator — Assistant professor of obstetrics and gynecology faculty of medicine Alazhar university Cairo